CLINICAL TRIAL: NCT02356939
Title: Efficacy Of A Removable Intraductal Stent In Duct-To-Duct Biliary Reconstruction To Prevent Biliary Complications In Liver Transplantation: A Randomized Controlled Trial
Brief Title: Removable Intraductal Stenting in Duct-to-duct Biliary Reconstruction in Liver Transplantation
Acronym: BILIDRAINT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interruption of the study for safety reasons at the decision of the sponsor
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P 130919
Record Dates: First submitted 2015-02-02; First posted 2015-02-06 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Transplantation, Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraductal stent (IST) (Experimental): For intervention : intraductal removable stent In the IST group, the surgeon will place the IST in the bile duct, which is a custom-made segment (2 cm) of a 8 French T-tube. The stent is inserted in the biliary duct without suture fixation.
  In the IST group, an endoscopic retrograde cholangio-pancreatography (ERCP) with sphincterotomy will be planned between the 4th and the 6th month post-transplantation.
  Interventions: Device: intraductal removable stent custom-made segment (2 cm)
- Without intraductal stent (no IST) (Experimental): For intervention : stent extraction by endoscopic retrograde cholangio-pancreatography (ERCP) Each center will perform its habitual postoperative follow up.
  Interventions: Procedure: stent extraction by ERCP

INTERVENTIONS:
Device: intraductal removable stent custom-made segment (2 cm) — : In the IST group, the surgeon will place the IST in the bile duct, which is a custom-made segment (2 cm) of a 8 French T-tube. The stent is inserted in the biliary duct without suture fixation.
  In order to minimize bias and to homogenize the technique, a short technical explanatory movie was realized by the promoter's team and edited on internet.
  In the IST group, an endoscopic retrograde cholangio-pancreatography (ERCP) with sphincterotomy will be planned between the 4th and the 5th month post-transplantation, requiring a short stay in hospital, a general anesthesia, clinical and biological tests including plasmatic lipase dosage at Day 1.
  Arms: Intraductal stent (IST)
Procedure: stent extraction by ERCP — stent extraction by endoscopic retrograde cholangio-pancreatography
  Arms: Without intraductal stent (no IST)

SUMMARY:
Randomized controlled trial including 7 French transplantation centers. Pre-inclusion of the patients is made when enlisted for liver transplantation (LT). Definitive inclusion and randomization is performed during LT, for patients undergoing a duct-to-duct biliary anastomosis with a graft bile duct diameter smaller than 7mm. In the intraductal stent tube group, a custom-made segment of a T-tube is placed into the bile duct, and removed endoscopically four to six months postoperative. The surgical technique is available on a movie during randomization on the website. The primary endpoint is the occurrence of biliary complications, including biliary fistulae and strictures, during six months of follow-up. Secondary evaluation criteria are the incidence of complications related to the stent placement and its extraction by endoscopy.

Discussion: Biliary complications following LT are significant causes of morbidity, retransplantation and eventually mortality. Although controversial, the use of a T-tube has been proven to be useless and even responsible for specific complications in many studies, including several randomized trials. However, several studies have identified a small bile duct diameter as a risk factor for biliary stenosis. A threshold of 7mm was found to be significantly associated to biliary stenosis. Our team published a preliminary study including 20 patients using a new technique of intraductal stenting. Only 4 complications were reported in the overall study population while no biliary complication occurred in the subgroup of patients who received a whole graft LT. Moreover, no technical failure and no procedure-related complications were noted before and during drain removal. Although intraductal stent tube in duct-to duct biliary anastomosis seems feasible and safe, a multicentric randomized controlled study is needed to validate it as a protective tool for biliary complications following LT.

DETAILED DESCRIPTION:
Comparative, multicentric, prospective, randomized non-blinded, two-groups study.

The follow-up is set at six months postoperative for a good screening of the majority of biliary complications.

The inclusion period is set at 3.5 years, for total study duration of 4 years. The patients' inclusion will be made in 7 liver transplantation centers in France.

Patients' inclusion will be performed in consultation at the moment of enlistment for LT, where they will be informed of the content, the benefits and risks of the study, and have to sign a written consent.

Definitive inclusion will be performed in operating room, during LT, and depends on fulfilling of the following "definitive inclusion criteria" (see above).

The randomization will be performed in operating room by the investigator and coordinated by the Clinical Research Unit of promoters' center (Saint Antoine Hospital, Paris), with a specific software accessible on the Internet.

In the IST group, the surgeon will place the IST in the bile duct, which is a custom-made segment (2 cm) of a 8 French T-tube with no side holes. The stent is inserted in the biliary duct without suture fixation.

In order to minimize bias and to homogenize the technique, a short technical explanatory movie will be realized by the promoter's team and distributed in each center.

Each center will perform its habitual postoperative follow up. Clinical, biological, and radiological exhaustive data will be collected at Day 1, Day 7, Day 15, Month 1, Month 3, Month 6.

A Magnetic Resonance Cholangiography (MRC) will be systematically performed at six months post LT.

In the IST group, an endoscopic retrograde cholangio-pancreatography (ERCP) with sphincterotomy will be planned between the 4th and the 5th month post-transplantation, requiring a short stay in hospital, a general anesthesia, clinical and biological tests including plasmatic lipase dosage at Day 1.

Every undesirable event will be immediately reported to the promoter for further investigation within its severity. Severe undesirable events will be previously defined.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for a liver transplantation
* Patients' written informed consent signed
* Patient with social coverage (excepting AME)

Exclusion criteria:

* Biliary reconstruction decided to be a hepaticojejunostomy for anatomical/biliary disease reason
* Non eligibility for liver transplantation:

  1. - Uncontrolled infectious process
  2. - Incompatible physical or mental state with the observance of the immunosuppressive drugs
  3. - Cardiopulmonary comorbidities severe / uncontrolled
  4. - Active alcohol intoxication or addiction
  5. - Pregnant or breastfeeding women (pregnancy test will be performed at baseline)
* Latex Allergy, polymer or rubber
* Patient participating in another interventional study about biliary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2015-04-03 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Incidence of biliary strictures and biliary fistulae within six months post-transplantation. | 6 months
  A biliary leakage is defined by the presence of bile in the abdominal drainage, and/or an intra-abdominal collection with bilious content requiring drainage.
  A biliary stenosis is defined by a size discrepancy between the two sides of the bile duct anastomosis on specific imaging (MR cholangiography, ERCP), associated to an upstream bile tract distention, with a clinical and biological cholestasis, after excluding other cholestasis causes (rejection, viral reactivation).

SECONDARY OUTCOMES:
Incidence of specific complications related to the IST and its extraction by endoscopy | 6 months
  Secondary endpoints are the incidence of specific complications related to the IST and its extraction by endoscopy: cholangitis, stent migration, extraction difficulties, acute pancreatitis, digestive perforation, hemorrhage.
Graft survival | 6 months
  Incidence of graft loss, i.e. retransplantation rate
Patient survival | 6 months
  Incidence of patient death

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SCATTON, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Olivier SOUBRANE, PU-PH, Study Director — Assistance Publique - Hôpitaux de Paris; Claire GOUMARD, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpétrière, Paris, France

REFERENCES:
- [Background] National Institutes of Health Consensus Development Conference Statement: liver transplantation--June 20-23, 1983. Hepatology. 1984 Jan-Feb;4(1 Suppl):107S-110S. No abstract available. PMID 6363254
- [Background] Consensus conference: Indications for Liver Transplantation, January 19 and 20, 2005, Lyon-Palais Des Congres: text of recommendations (long version). Liver Transpl. 2006 Jun;12(6):998-1011. doi: 10.1002/lt.20765. No abstract available. PMID 16721776
- [Background] Neuhaus P, Blumhardt G, Bechstein WO, Steffen R, Platz KP, Keck H. Technique and results of biliary reconstruction using side-to-side choledochocholedochostomy in 300 orthotopic liver transplants. Ann Surg. 1994 Apr;219(4):426-34. doi: 10.1097/00000658-199404000-00014. PMID 8161269
- [Background] Akamatsu N, Sugawara Y, Hashimoto D. Biliary reconstruction, its complications and management of biliary complications after adult liver transplantation: a systematic review of the incidence, risk factors and outcome. Transpl Int. 2011 Apr;24(4):379-92. doi: 10.1111/j.1432-2277.2010.01202.x. Epub 2010 Dec 10. PMID 21143651
- [Background] Roberts MS, Angus DC, Bryce CL, Valenta Z, Weissfeld L. Survival after liver transplantation in the United States: a disease-specific analysis of the UNOS database. Liver Transpl. 2004 Jul;10(7):886-97. doi: 10.1002/lt.20137. PMID 15237373
- [Background] Jain A, Reyes J, Kashyap R, Dodson SF, Demetris AJ, Ruppert K, Abu-Elmagd K, Marsh W, Madariaga J, Mazariegos G, Geller D, Bonham CA, Gayowski T, Cacciarelli T, Fontes P, Starzl TE, Fung JJ. Long-term survival after liver transplantation in 4,000 consecutive patients at a single center. Ann Surg. 2000 Oct;232(4):490-500. doi: 10.1097/00000658-200010000-00004. PMID 10998647
- [Background] Sharma S, Gurakar A, Jabbour N. Biliary strictures following liver transplantation: past, present and preventive strategies. Liver Transpl. 2008 Jun;14(6):759-69. doi: 10.1002/lt.21509. PMID 18508368
- [Background] Duailibi DF, Ribeiro MA Jr. Biliary complications following deceased and living donor liver transplantation: a review. Transplant Proc. 2010 Mar;42(2):517-20. doi: 10.1016/j.transproceed.2010.01.017. PMID 20304182
- [Background] Park JB, Kwon CH, Choi GS, Chun JM, Jung GO, Kim SJ, Joh JW, Lee SK. Prolonged cold ischemic time is a risk factor for biliary strictures in duct-to-duct biliary reconstruction in living donor liver transplantation. Transplantation. 2008 Dec 15;86(11):1536-42. doi: 10.1097/TP.0b013e31818b2316. PMID 19077886
- [Background] Marubashi S, Dono K, Nagano H, Kobayashi S, Takeda Y, Umeshita K, Monden M, Doki Y, Mori M. Biliary reconstruction in living donor liver transplantation: technical invention and risk factor analysis for anastomotic stricture. Transplantation. 2009 Nov 15;88(9):1123-30. doi: 10.1097/TP.0b013e3181ba184a. PMID 19898209
- [Background] Hwang S, Lee SG, Sung KB, Park KM, Kim KH, Ahn CS, Lee YJ, Lee SK, Hwang GS, Moon DB, Ha TY, Kim DS, Jung JP, Song GW. Long-term incidence, risk factors, and management of biliary complications after adult living donor liver transplantation. Liver Transpl. 2006 May;12(5):831-8. doi: 10.1002/lt.20693. PMID 16528711
- [Background] Shaked A. Use of T tube in liver transplantation. Liver Transpl Surg. 1997 Sep;3(5 Suppl 1):S22-3. No abstract available. PMID 9377769
- [Background] Rolles K, Dawson K, Novell R, Hayter B, Davidson B, Burroughs A. Biliary anastomosis after liver transplantation does not benefit from T tube splintage. Transplantation. 1994 Feb;57(3):402-4. doi: 10.1097/00007890-199402150-00015. PMID 8108875
- [Background] Ben-Ari Z, Neville L, Davidson B, Rolles K, Burroughs AK. Infection rates with and without T-tube splintage of common bile duct anastomosis in liver transplantation. Transpl Int. 1998;11(2):123-6. doi: 10.1007/s001470050115. PMID 9561678
- [Background] Vougas V, Rela M, Gane E, Muiesan P, Melendez HV, Williams R, Heaton ND. A prospective randomised trial of bile duct reconstruction at liver transplantation: T tube or no T tube? Transpl Int. 1996;9(4):392-5. doi: 10.1007/BF00335701. PMID 8819276
- [Background] Scatton O, Meunier B, Cherqui D, Boillot O, Sauvanet A, Boudjema K, Launois B, Fagniez PL, Belghiti J, Wolff P, Houssin D, Soubrane O. Randomized trial of choledochocholedochostomy with or without a T tube in orthotopic liver transplantation. Ann Surg. 2001 Mar;233(3):432-7. doi: 10.1097/00000658-200103000-00019. PMID 11224633
- [Background] Weiss S, Schmidt SC, Ulrich F, Pascher A, Schumacher G, Stockmann M, Puhl G, Guckelberger O, Neumann UP, Pratschke J, Neuhaus P. Biliary reconstruction using a side-to-side choledochocholedochostomy with or without T-tube in deceased donor liver transplantation: a prospective randomized trial. Ann Surg. 2009 Nov;250(5):766-71. doi: 10.1097/SLA.0b013e3181bd920a. PMID 19809299
- [Background] Zalinski S, Soubrane O, Scatton O. Reducing biliary morbidity in full graft deceased donor liver transplantation: is it really a matter of T-tube? Ann Surg. 2010 Sep;252(3):570-1; author reply 571-2. doi: 10.1097/SLA.0b013e3181f07a6b. No abstract available. PMID 20739862
- [Background] Lopez-Andujar R, Oron EM, Carregnato AF, Suarez FV, Herraiz AM, Rodriguez FS, Carbo JJ, Ibars EP, Sos JE, Suarez AR, Castillo MP, Pallardo JM, De Juan Burgueno M. T-tube or no T-tube in cadaveric orthotopic liver transplantation: the eternal dilemma: results of a prospective and randomized clinical trial. Ann Surg. 2013 Jul;258(1):21-9. doi: 10.1097/SLA.0b013e318286e0a0. PMID 23426348
- [Background] Sherman S, Jamidar P, Shaked A, Kendall BJ, Goldstein LI, Busuttil RW. Biliary tract complications after orthotopic liver transplantation. Endoscopic approach to diagnosis and therapy. Transplantation. 1995 Sep 15;60(5):467-70. doi: 10.1097/00007890-199509000-00011. PMID 7676495
- [Background] Ostroff JW. Post-transplant biliary problems. Gastrointest Endosc Clin N Am. 2001 Jan;11(1):163-83. PMID 11175980
- [Background] Vandenbroucke F, Plasse M, Dagenais M, Lapointe R, Letourneau R, Roy A. Treatment of post liver transplantation bile duct stricture with self-expandable metallic stent. HPB (Oxford). 2006;8(3):202-5. doi: 10.1080/13651820500501800. PMID 18333277
- [Background] Chaput U, Scatton O, Bichard P, Ponchon T, Chryssostalis A, Gaudric M, Mangialavori L, Duchmann JC, Massault PP, Conti F, Calmus Y, Chaussade S, Soubrane O, Prat F. Temporary placement of partially covered self-expandable metal stents for anastomotic biliary strictures after liver transplantation: a prospective, multicenter study. Gastrointest Endosc. 2010 Dec;72(6):1167-74. doi: 10.1016/j.gie.2010.08.016. PMID 20970790
- [Background] Farhat S, Bourrier A, Gaudric M, Dousset B, Scatton O, Chaussade S, Prat F. Endoscopic treatment of biliary fistulas after complex liver resection. Ann Surg. 2011 Jan;253(1):88-93. doi: 10.1097/SLA.0b013e3181f9b9f0. PMID 21233609
- [Background] Tranchart H, Zalinski S, Sepulveda A, Chirica M, Prat F, Soubrane O, Scatton O. Removable intraductal stenting in duct-to-duct biliary reconstruction in liver transplantation. Transpl Int. 2012 Jan;25(1):19-24. doi: 10.1111/j.1432-2277.2011.01339.x. Epub 2011 Sep 29. PMID 21954951
- [Background] Cotton PB, Garrow DA, Gallagher J, Romagnuolo J. Risk factors for complications after ERCP: a multivariate analysis of 11,497 procedures over 12 years. Gastrointest Endosc. 2009 Jul;70(1):80-8. doi: 10.1016/j.gie.2008.10.039. Epub 2009 Mar 14. PMID 19286178
- [Background] Gastaca M. Biliary complications after orthotopic liver transplantation: a review of incidence and risk factors. Transplant Proc. 2012 Jul-Aug;44(6):1545-9. doi: 10.1016/j.transproceed.2012.05.008. PMID 22841209
- [Background] CATTELL RB, BRAASCH JW. An eveluation of the long T-tube. Ann Surg. 1961 Aug;154(2):252-4. doi: 10.1097/00000658-196108000-00009. No abstract available. PMID 13691630
- [Derived] Goumard C, Boleslawski E, Brustia R, Dondero F, Herrero A, Lesurtel M, Barbier L, Lecolle K, Soubrane O, Bouyabrine H, Mabrut JY, Salame E, Cachanado M, Simon T, Scatton O. Duct-to-duct biliary reconstruction with or without an intraductal removable stent in liver transplantation: The BILIDRAIN-T multicentric randomised trial. JHEP Rep. 2022 Jul 6;4(10):100530. doi: 10.1016/j.jhepr.2022.100530. eCollection 2022 Oct. PMID 36082313
- [Derived] Goumard C, Cachanado M, Herrero A, Rousseau G, Dondero F, Compagnon P, Boleslawski E, Mabrut JY, Salame E, Soubrane O, Simon T, Scatton O. Biliary reconstruction with or without an intraductal removable stent in liver transplantation: study protocol for a randomized controlled trial. Trials. 2015 Dec 30;16:598. doi: 10.1186/s13063-015-1139-6. PMID 26719017